CLINICAL TRIAL: NCT06089772
Title: A Comparison Of The Effects Of High-Velocity Low-Amplitude (Hvla) Manipulation And Myofascial Release Technique On Performance In Healthy Individuals With Sacroiliac Joint Dysfunction
Brief Title: Manipulation and Myofascial Techniques On Sacroiliac Joint Dysfunction
Acronym: HVLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alanya Alaaddin Keykubat University (Other)
Responsible Party: Principal Investigator, Ayça Araci, PHD, Physiotherapist, Head of Physiotherapy and Rehabilitation Department, Alanya Alaaddin Keykubat University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 61351342
Record Dates: First submitted 2023-10-03; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Manipulation, Psychologic; Pain; Performance Anxiety; Participation, Patient; Physiotherapists
MeSH Terms: conditions — Pain; Patient Participation

STUDY DESIGN:
Intervention Model Description: The groups determined as randomly into the four groups. Group I (n=14) received HVLA spinal manipulation, Group II (n=14) underwent foam roller stretching, Group III (n=14) received a combination of HVLA spinal manipulation and foam roller stretching, and Group IV (n=14) underwent sham manipulation as the control group. Measures were measured before the acute intervention and right after the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group I (Experimental): Group I (n=14) received HVLA spinal manipulation
  Interventions: Other: Comparing to Manipulation and Myofascial Release Techniques
- Group II (Active Comparator): Group II (n=14) underwent foam roller stretching,
  Interventions: Other: Comparing to Manipulation and Myofascial Release Techniques
- Group III (Active Comparator): Group III (n=14) received a combination of HVLA spinal manipulation and foam roller stretching,
  Interventions: Other: Comparing to Manipulation and Myofascial Release Techniques
- Group IV (Sham Comparator): Group IV (n=14) underwent sham manipulation as the control group
  Interventions: Other: Comparing to Manipulation and Myofascial Release Techniques

INTERVENTIONS:
Other: Comparing to Manipulation and Myofascial Release Techniques — Randomized Controlled Trials

SUMMARY:
Aimed to compare the effects of High-Velocity Low-Amplitude (HVLA) manipulation and myofascial release techniques on performance in healthy individuals with sacroiliac joint dysfunction.

DETAILED DESCRIPTION:
Aim: aimed to compare the effects of High-Velocity Low-Amplitude (HVLA) manipulation and myofascial release techniques on performance in healthy individuals with sacroiliac joint dysfunction. Design: Randomized control trial. Setting: University physiotherapy clinic. Participiants: Participants aged 18-45 years with confirmed Dysfunction by six clinical Sacroiliac Joint diagnostic tests. Intervention: The groups determined as randomly into the four groups. Group I (n=14) received HVLA spinal manipulation, Group II (n=14) underwent foam roller stretching, Group III (n=14) received a combination of HVLA spinal manipulation and foam roller stretching, and Group IV (n=14) underwent sham manipulation as the control group. Measures were measured before the acute intervention and right after the intervention. Outcomes: Prior to the interventions, participants were evaluated using the Visual Analog Scale (VAS) for pain assessment, the Baseline Sit and Reach test for flexibility assessment, the Optojump Next system (Via Stradivari, Bolzano) for vertical jump performance and multiple jump tests, and the MicroFet2 digital hand dynamometer (United States, Utah) for muscle strength measurement. Results: The study groups showed statistically significant improvements in performance parameters compared to the control group (p<0.05). Pre-treatment and post-treatment performance parameters and pain values were statistically significant in both groups (p<0.05). While performance improvements were observed in all four groups, the highest changes were generally observed in the HVLA + Myofascial release group. Conclusion: Considering the overall results, the combined use of HVLA and Myofascial release in the treatment protocol is recommended.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer
2. Being between the ages of 18-45,
3. Not to have any psychological, neurological, orthopedic and rheumatic disorders,
4. Not having any other musculoskeletal pathology affecting the lower extremities,
5. Not having undergone spine and/or lower extremity surgery,
6. Those with mechanical sacroiliac joint pain,
7. Patients in whom at least 3 out of 6 provocation tests showing sacroiliac joint dysfunction and validity-reliability studies were positive: 1. Distraction, 2. Compression, 3. Gaenslen, 4. Posterior friction test, 5. Sacral thrust, 6. Faber (8) Individuals with sacroiliac pain at least 3 points on the VAS in the last 1 month 11

Exclusion Criteria:

1. Being under the age of 18 and over the age of 45,
2. Having any psychological, neurological, orthopedic and rheumatic disorders,
3. Pregnancy and suspicion of pregnancy,
4. Having active malignancies,
5. Having an active infection,
6. Injection and operation of the sacroiliac joint in the last 3 months,
7. Having drug or substance addiction,
8. Central vascular/neurological conditions

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Baseline - right after the intervention
  Pain Level Measurement - When reading the VAS, the position of the respondent's cross is generally assigned a score between 0 and 100. If documented in paper form, the scores can then be simply transferred to a 100-value scale using a millimeter tape measure. The division into hundredths is considered sufficiently sensitive.
Baseline Sit and Reach Test | Baseline - right after the intervention
  Flexibility - A standard SR box was placed on the floor by placing tape at a right angle to the 38 cm mark. The participants sat on the floor with shoes on and fully extended one leg so that the sole of the foot was flat against the end of the box. They then extended their arms forward, placing one hand on top of the other. With palms down, they reached forward, sliding hands along the measuring scale as far as possible without bending the knee of the extended leg. Throughout testing, the physiotherapist (NU) heel remained at the 45 cm mark.
The Optojump Next system (Via Stradivari, Bolzano) for vertical jump performance | Baseline - right after the intervention
  Participants were positioned in a mini squat with arms held back, starting from the initial position. Participants were instructed to perform 3 consecutive vertical jumps, lifting their arms upward from the front. The average of the three measurements was calculated for jump performance and recorded in centimeters. Glatthorn et al., (2011) reported an interrater reliability ICC value between 0.997 and 0.998 for the Optojump Next device in estimating vertical jump height
The Optojump Next system (Via Stradivari, Bolzano) for multiple jump tests, | Baseline - right after the intervention
  Upon the practitioner's 'start' command, participants continuously jumped vertically for 15 seconds, maintaining their knees extended and hands free. At the end of the test, using the computer and camera connected to the measurement device, values (jump count, contact time, airborne time, height, power, step) were recorded
MicroFet2 digital hand dynamometer | Baseline - right after the intervention
  Muscle strength measurement was performed for the hamstring, gastrocnemius, and soleus muscles. For muscle strength measurement, the MicroFet2 digital handheld dynamometer (United States, Utah) was used 17. To ensure maximum isometric contraction for each muscle group, the application was repeated 3 times, with each contraction held for 5 seconds, and there were 15-second breaks between repetitions 18,19Participants were briefed about the procedures and were given 2 practice trials. After the practice trials, a 1-minute break was given before the actual measurements began.

CONTACTS AND LOCATIONS:
Locations (1):
- Ayça ARACI, Alanya, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided